CLINICAL TRIAL: NCT05915884
Title: Investigation of the Triglyceride/Glucose Index in Diabetic Patients Using SGLT-2 Inhibitor
Brief Title: The Triglyceride/Glucose Index and SGLT-2 Inhibitors
Status: Completed | Type: Observational
Sponsor: Samsun Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Duriye Sila Karagoz Ozen, MD,Internal Medicine Specialist, Samsun Education and Research Hospital
Other Study IDs: 1
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Metabolic Disease; Diabetes
Keywords: SGLT-2 inhibitor; triglyceride index
MeSH Terms: conditions — Metabolic Diseases; Diabetes Mellitus | interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type 2 diabetic patients using SGLT-2 inhibitors: The data of all patients who applied to Samsun Training and Research Hospital Internal Medicine outpatient clinic for 12 months in 2022 and were started on SGLT-2 inhibitor will be examined. According to the inclusion and exclusion criteria, the patients will be evaluated and the data of the patients admitted to the study will be analyzed. The triglyceride glucose index of the patients before starting the SGLT-2 treatment and the triglyceride glucose index at the end of 3 months of treatment will be calculated by the researchers using the data in the system. No additional blood tests or laboratory analyses will be performed on the patients.
  Interventions: Other: SGLT-2 inhibitors

INTERVENTIONS:
Other: SGLT-2 inhibitors — This study is an observational study. It is not planned to do an interventional activity.

SUMMARY:
This study was designed to evaluate the change in triglyceride glucose index, one of the atherosclerotic markers, in patients with type 2 DM followed in the Internal Medicine Clinic of Samsun University, Samsun Training, and Research Hospital.

Methods: The data of the patients who were followed up for at least 3 months by making a retrospective file review will be recorded and analyzed. It is planned to start the study following the ethics committee's approval.

DETAILED DESCRIPTION:
The data of all patients who applied to Samsun Training and Research Hospital Internal Medicine outpatient clinic for 12 months in 2022 and were started on SGLT-2 inhibitor will be examined. According to the inclusion and exclusion criteria stated below, the patients will be evaluated and the data of the patients admitted to the study will be analyzed. The triglyceride glucose index of the patients before starting the SGLT-2 injection and the trig/glucose index at the end of 3 months of treatment will be calculated by the researchers using the data in the system. No additional blood tests or laboratory analyses will be performed on the patients. Triglyceride, glucose, and glycosylated hemoglobin values were checked at the beginning of the treatment and at the 3rd-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 DM
* Age >18 years old
* Dapagliflozin 10 mg or empagliflozin 10 mg or 25 mg
* 3 months follow-up period

Exclusion Criteria:

* Type 1 diabetes
* Gestational diabetes
* Age < 18 years old
* Insufficient or missed laboratory test results
* Medical treatment for dyslipidemia
* Hypothyroidism

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a diagnosis of type 2 Diabetes Mellitus who applied to Samsun Training and Research Hospital Internal Medicine outpatient clinic for 12 months in 2022 and were started on SGLT-2 inhibitor will be examined. According to the inclusion and exclusion criteria stated above, the patients will be evaluated and the data of the patients admitted to the study will be analyzed.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2023-06-10 (Actual); Primary Completion 2023-10-28 (Actual); Study Completion 2024-01-28 (Actual)

PRIMARY OUTCOMES:
Change in triglyceride index | 3 months
  Decreased triglyceride index among patients using SGLT-2 inhibitors.

CONTACTS AND LOCATIONS:
Overall Officials: DÜRİYE SILA KARAGÖZ ÖZEN, Principal Investigator — Samsun Education and Research Hospital
Locations (1):
- Samsun Education and Research Hospital, Samsun, İlkadım, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided